CLINICAL TRIAL: NCT01144676
Title: A Double-Blind, Randomised, Placebo-Controlled Pharmacokinetic and Safety Trial in Healthy HIV-Negative Women to Assess the Delivery of Dapivirine From a Matrix Vaginal Ring and to Evaluate the Safety of a Matrix Vaginal Ring Containing 25 MG of Dapivirine
Brief Title: A Safety Study to Assess the Delivery of Dapivirine From a Matrix Vaginal Ring
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Annalene Nel, MBChB, PhD, IPM
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IPM 013
Record Dates: First submitted 2010-06-10; First posted 2010-06-15 (Estimated); Last update posted 2010-10-06 (Estimated); Status verified 2010-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Dapivirine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A1: Dapivirine Vaginal Ring (Experimental)
  Interventions: Drug: dapivirine
- Group A2: Placebo Vaginal Ring (Placebo Comparator)
  Interventions: Drug: placebo
- Group B1: Dapivirine Vaginal Ring (Experimental)
  Interventions: Drug: dapivirine
- Group B2: Placebo Vaginal Ring (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: dapivirine — 25mg dapivirine per ring.
  The first vaginal ring will be removed on Day 28, and a new vaginal ring will be reinserted after 3 days, on day 31, for another 28 days.
  Arms: Group A1: Dapivirine Vaginal Ring
Drug: placebo — The first vaginal ring will be removed on Day 28, and a new vaginal ring will be reinserted after 3 days, on day 31, for another 28 days.
  Arms: Group A2: Placebo Vaginal Ring
Drug: dapivirine — 25mg dapivirine per ring.
  The first vaginal ring will be removed on day 35 and the new vaginal ring will be reinserted after 3 days, on day 38, for another 21 days. A third vaginal ring will be inserted immediately following removal of second ring on Day 59 and will be worn for 24 hours.
  Arms: Group B1: Dapivirine Vaginal Ring
Drug: placebo — The first vaginal ring will be removed on day 35 and the new vaginal ring will be reinserted after 3 days, on day 38, for another 21 days. A third vaginal ring will be inserted immediately following removal of second ring on Day 59 and will be worn for 24 hours.
  Arms: Group B2: Placebo Vaginal Ring

SUMMARY:
The proposed study is a single-center, double-blind, randomised, placebo-controlled trial to evaluate the delivery of dapivirine from matrix vaginal rings over a 56 and 57 day period and to assess the safety as compared to placebo vaginal rings in 48 healthy, HIV-negative, sexually active women.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 and ≤40 years of age who can give written informed consent;
* Available for all visits and consent to follow all procedures scheduled for the trial;
* Healthy and self-reported sexually active (defined as an average of one penetrative penile vaginal coital act per month for the 3 months prior to enrolment);
* Be on a stable form of contraception, defined as:

  * A stable oral contraceptive regimen for at least 2 months prior to enrolment, OR,
  * Transdermal contraceptive patch for at least 3 months prior to enrolment, OR,
  * Long-acting progestins for at least 6 months prior to enrolment, OR,
  * An IUD inserted (with no vaginal or gynaecological complaints associated with its use) at least 3 months prior to enrolment, OR,
  * Have undergone surgical sterilization at least 3 months prior to enrolment;
* In the absence of the use of exogenous hormone(s), have a self-reported regular menstrual cycle, defined as having a minimum of 21 days and a maximum of 35 days between menses;
* Upon pelvic examination and colposcopy at the time of enrolment, the cervix and vagina appear normal as determined by the Investigator;
* Asymptomatic for genital infections at the time of enrolment (if a woman is diagnosed with any treatable STI, either syndromically or by laboratory test at the time of screening, she must receive treatment at least 2 weeks prior to enrolment);
* Willing to refrain from the use of vaginal products or objects including, female condoms, cotton wool, rags, diaphragms, cervical caps (or any other vaginal barrier method), douches, lubricants, vibrators/dildos, and drying agents for 14 days prior to enrolment and for the duration of the trial. Tampon use will be permitted;
* Willing to use oral contraceptives to avoid menstruation, if necessary while taking part in this trial;
* Documentation of no abnormality on Pap test, including grossly bloody smear, within 90 days prior to screening;
* Willing to refrain from participation in any other research trial for the duration of this trial;
* Willing to provide adequate locator information for trial retention purposes and be reachable per local standard procedures [e.g., by home visit or telephone; or via family or close neighbour contacts (confidentiality to be maintained)];
* Willing to agree to abstain from all the following criteria for a total of 2 days (48 hours) prior to each trial visit, as well as for a total of 3 days (72 hours) after the biopsy procedure:

  * Vaginal intercourse
  * Oral contact with her genitalia
* Hepatitis B and C negative at the time of enrolment.

Exclusion Criteria:

* Currently pregnant or having had their last pregnancy outcome within 3 months prior to screening;
* Currently breast-feeding;
* Currently or within two months of participation in any other clinical research trial involving investigational or marketed products prior to screening;
* Untreated symptomatic urogenital infections, e.g., urinary tract or other sexually transmitted infections, or other gynaecological conditions such as vaginal itching, pain, or discharge, within 2 weeks prior to enrolment;
* Presence of any abnormal clinically significant physical finding on the vulva, vaginal walls or cervix during pelvic examination and/or colposcopy at pre-enrolment;
* History of urogenital or uterine prolapse, undiagnosed vaginal bleeding, urethral obstruction, incontinence or urge incontinence;
* Current vulvar or vaginal symptoms / abnormalities that could influence the trial results;
* Pap test result that requires cryotherapy, biopsy, treatment (other than for infection); or further evaluation [this includes any findings of atypical squamous cells of undetermined significance (ASCUS)];
* Symptomatic genital HSV infection or a history of genital herpetic infection;
* Any Grade 2, 3 or 4 haematology, chemistry or urinalysis laboratory abnormality at baseline (screening) according to the DAIDS Table for Grading Adverse Events (NOTE: This table can be found at: http://rcc.tech-res.com/safetyandpharmacovigilance;and a standardized version will be provided to the research centre in the Study Operations Manual);
* Unexplained, abnormal bleeding per vagina during or following vaginal intercourse, or gynaecologic surgery within 90 days prior to enrolment;
* Any history of anaphylaxis or severe allergy resulting in angioedema; or a history of sensitivity/allergy to latex or silicone;
* Any serious acute, chronic or progressive disease (e.g., any known history of neoplasm, cancer, diabetes, cardiac disease, autoimmune disease, HIV, AIDS, or blood dyscrasias), or signs of cardiac disease, renal failure, or severe malnutrition;
* Have undergone a hysterectomy;
* Any condition(s) that, in the opinion of the Investigator, might interfere with adherence to trial requirements or evaluation of the trial objectives.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety: To assess the safety of the dapivirine vaginal ring, the endpoint was the proportion of women in four vaginal ring regimens on dapivirine or placebo ring experiencing specific, protocol-defined safety events during the study (see description) | 56/57 days
  * Mucosal abnormalities (as defined in the CONRAD/WHO manual) visible during naked eye examination and/or colposcopy;
  * Abnormal vaginal pH and/or abnormal vaginal flora during the course of the trial.
  * Positive diagnostic tests for trichomonas, gonorrhoea and/or chlamydia;
  * At least one adverse event during the 12-week trial period;
  * Any laboratory abnormalities on haematology, electrolytes, liver function, and renal function.
Pharmacokinetics: To examine local and systemic pharmacokinetics of dapivirine concentrations delivered by the vaginal rings, measured in plasma, vaginal fluids and cervical tissue during the trial period | 56/57 days

CONTACTS AND LOCATIONS:
Overall Officials: Annelene Nel, PhD, Study Director — Beijing Immupeutics Medicine Technology Limited
Locations (1):
- SGS Life Science Services, Antwerp, Flanders, Belgium